CLINICAL TRIAL: NCT00005128
Title: Lipid Research Clinics Population Studies
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 907
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2004-04

CONDITIONS: Cardiovascular Diseases; Atherosclerosis; Coronary Disease; Heart Diseases; Hyperlipoproteinemia
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Coronary Disease; Heart Diseases; Hyperlipoproteinemias

SUMMARY:
To conduct epidemiologic surveys of the distribution, causes, and consequences of the dyslipoproteinemias. The Population Studies include the Prevalence Study, the Family Study, and the Mortality Follow-up Study and shared the same general population base.

DETAILED DESCRIPTION:
BACKGROUND:

The Lipid Research Clinics program was created in 1971. The objectives were to evaluate the then current techniques for diagnosis of hyperlipoproteinemia; to acquire data across all age groups on the prevalence of different types of hyperlipoproteinemia, particularly genetically determined forms; to collect high quality data on the prevalence and incidence of atherosclerosis in different patterns of hyperlipoproteinemia; and to improve methods for detection, diagnosis, and medical care of coronary heart disease. The program consisted of the Population Studies and the Coronary Primary Prevention Trial. The coronary primary prevention trial is described under Clinical Trials in the database.

As a result of the establishment of the U.S.-U.S.S.R. Joint Program in Cardiovascular Diseases in 1972, lipid research clinics were established in Moscow and Leningrad in 1974. The U.S.S.R. component of this collaborative research consisted of two Prevalence Studies and a Follow-up Study, all of which closely followed the U.S. Lipid Research Clinics Prevalence Study protocol.

DESIGN NARRATIVE:

Prevalence Study:

The Prevalence Study was initiated in 1972 to determine the prevalence of different types of dyslipoproteinemias at ten North American Lipid Research Clinics. The Prevalence Study consisted of two screens designated as Visit 1 and Visit 2, and was conducted according to a standardized protocol in well-defined target populations. Data collection began in 1972 and ended in 1976. The median time between the two screens was 96 days. The objectives of Visit 1 were: to provide estimates of the prevalence of dyslipidemia in specified populations; to investigate the distribution of cholesterol and triglyceride; and to select participants for Visit 2. A total of 60,502 eligible participants were screened at visit 1. A 15 percent random sample (N=9,107) of all Visit 1 participants who had elevated lipids (N=6,882) or were taking lipid-altering medication (N=346) were asked to return for the Lipid Research Clinics Population Studies Visit 2 screen. The three groups of 16,335 participants represented approximately 25 percent of all subject screened at Visit 1. The objectives of Visit 2 were: to identify participants with primary or secondary dyslipoproteinemia; to determine the prevalence of lipid and lipoprotein patterns and their associations with coronary heart disease, other vascular diseases, and other risk factors for coronary heart disease; and to determine the relationships between lipids and lipoprotein patterns and selected nutritional, physiologic, and sociodemographic variables such as education and occupation of head of household, smoking, blood pressure, height, weight, triceps skinfold, Quetelet index, and sex hormone usage by females. Visit 2 procedures included an interview, a physical examination, an ECG, clinical chemistries, and one-day dietary recall.

Family Study:

The Family Study provided data on the relationship of familial and genetic attributes to plasma lipids and lipoproteins. A sample of all participants in Visit 2 of the Prevalence Study was chosen to participate as probands. Basic demographic information was collected and plasma lipids and lipoproteins were measured on all first-degree relatives and probands. The Family Study was initiated in 1975 and data collection was completed in 1978.

Follow-Up Study:

The Follow-up Study, initiated in 1977, was designed to relate the baseline observation made in 1972-1976 to total and cause-specific mortality. The study assessed the risk factor status of plasma triglycerides, HDL cholesterol and exercise electrocardiography for cardiovascular disease mortality in general, and coronary heart disease in particular. Follow-up baseline measurements included lipid and other clinical chemistries, one-day dietary recalls, medication histories and physical examinations. Assessments were also made of the relationships of estrogen use in women to subsequent cardiovascular disease, coronary heart disease, and cancer mortality and of the relationships of lipids and lipoprotein levels to site-specific cancer, as well as the relationship of retinol levels to cancer mortality.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1972-07; Study Completion 1994-12

REFERENCES:
- [Background] Ahmed S, Lippel K, Bachorik PS, Muesing R, Weidman S, Winn C. External quality control survey of triglyceride (triacylglycerol) analyses performed by 12 lipid research clinics. Clin Chem. 1979 Jun;25(6):880-8. No abstract available. PMID 445825
- [Background] Bachorik PS, Wood PD, Williams J, Kuchmak M, Ahmed S, Lippel K, Albers J. Automated determination of total plasma cholesterol: a serum calibration technique. Clin Chim Acta. 1979 Aug 15;96(1-2):145-53. doi: 10.1016/0009-8981(79)90064-0. PMID 476955
- [Background] Kuba K, Lippel K, Frantz ID Jr. Four electrophoretic methods compared for diagnosis of type III hyperlipoproteinemia. Clin Chem. 1979 Aug;25(8):1471-5. PMID 222508
- [Background] Wood PD, Bachorik PS, Albers JJ, Stewart CC, Winn C, Lippel K. Effects of sample aging on total cholesterol values determined by the automated ferric chloride-sulfuric acid and Liebermann-Burchard procedures. Clin Chem. 1980 Apr;26(5):592-7. PMID 7261302
- [Background] Warnick GR, Albers JJ, Bachorik PS, Turner JD, Garcia C, Breckinridge C, Kuba K, McNeely S, Hillerman G, King P, Muesing R, Most B, Lippel K. Multilaboratory evaluation of an ultrafiltration procedure for high density lipoprotein cholesterol quantification in turbid heparin-manganese supernates. J Lipid Res. 1981 Aug;22(6):1015-20. PMID 7276749
- [Background] Bachorik PS, Most B, Lippel K, Albers JJ, Wood PD. Plasma lipoprotein analysis: relative precision of total cholesterol and lipoprotein-cholesterol measurements in 12 lipid-research-clinics laboratories. Clin Chem. 1981 Jul;27(7):1217-22. No abstract available. PMID 7237787
- [Background] Williams OD, Heiss G., Beaglehole R, Dennis B, Bazzarre T, and Tyroler HA: Hyperlipidemia and Nutrition - Data Base and Trends. Atherosclerosis Reviews 7:145-156, 1980
- [Background] Morrison JA, Khoury P, Laskarzewski P, Gartside P, Moore M, Heiss G, Glueck CJ. Hyperalphalipoproteinemia in hypercholesterolemic adults and children. Trans Assoc Am Physicians. 1980;93:230-43. PMID 7245576
- [Background] Christensen B, Glueck C, Kwiterovich P, Degroot I, Chase G, Heiss G, Mowery R, Tamir I, Rifkind B. Plasma cholesterol and triglyceride distributions in 13,665 children and adolescents: the Prevalence Study of the Lipid Research Clinics Program. Pediatr Res. 1980 Mar;14(3):194-202. doi: 10.1203/00006450-198003000-00004. PMID 6966785
- [Background] Tamir I, Heiss G, Glueck CJ, Christensen B, Kwiterovich P, Rifkind BM. Lipid and lipoprotein distributions in white children ages 6-19 yr. The Lipid Research Clinics Program Prevalence Study. J Chronic Dis. 1981;34(1):27-39. doi: 10.1016/0021-9681(81)90079-5. No abstract available. PMID 7451637
- [Background] Wallace RB, Lynch CF, Pomrehn PR, Criqui MH, Heiss G. Alcohol and hypertension: epidemiologic and experimental considerations. The Lipid Research Clinics Program. Circulation. 1981 Sep;64(3 Pt 2):III 41-7. PMID 7020983
- [Background] Glueck CJ, Heiss G, Morrison JA, Khoury P, Moore M. Alcohol intake, cigarette smoking and plasma lipids and lipoproteins in 12--19-year-old children. The Collaborative Lipid Research Clinics Prevalence Study. Circulation. 1981 Sep;64(3 Pt 2):III 48-56. PMID 7020984
- [Background] Gordon T, Ernst N, Fisher M, Rifkind BM. Alcohol and high-density lipoprotein cholesterol. Circulation. 1981 Sep;64(3 Pt 2):III 63-7. PMID 7020986
- [Background] Criqui MH, Wallace RB, Mishkel M, Barrett-Connor E, Heiss G. Alcohol consumption and blood pressure. The lipid research clinics prevalence study. Hypertension. 1981 Sep-Oct;3(5):557-65. doi: 10.1161/01.hyp.3.5.557. PMID 7298110
- [Background] Hunninghake D, Wallace RB, Reiland S, Barrett-Connor E, Wahl P, Hoover J, Heiss G. Alterations of plasma lipid and lipoprotein levels associated with benzodiazepine use--the LRC Program Prevalence Study. Atherosclerosis. 1981 Oct;40(2):159-65. doi: 10.1016/0021-9150(81)90034-4. PMID 6118165
- [Background] Wallace RB, Barrett-Connor E, Criqui M, Wahl P, Hoover J, Hunninghake D, Heiss G. Alteration in blood pressures associated with combined alcohol and oral contraceptive use-the lipid research clinics prevalence study. J Chronic Dis. 1982;35(4):251-7. doi: 10.1016/0021-9681(82)90081-9. PMID 7061681
- [Background] Cowan LD, Wallace RB, Barrett-Connor E, Hunninghake D, Pomrehn P, Wahl P, Heiss G. Alterations in clinical chemistry measures associated with oral contraceptive and estrogen use: the Lipid Research Clinics Program Prevalence Study. J Reprod Med. 1982 May;27(5):275-82. PMID 7108863
- [Background] Kwiterovich PO Jr, Heiss G, Johnson N, Chase GA, Tamir I, Rifkind B. Assessment of plasma total cholesterol as a test to detect elevated low density (beta) lipoprotein cholesterol levels (type IIa hyperlipoproteinemia) in young subjects from a population-based sample. Am J Epidemiol. 1982 Feb;115(2):192-204. doi: 10.1093/oxfordjournals.aje.a113291. PMID 7058778
- [Background] Criqui MH, Mebane I, Wallace RB, Heiss G, Holdbrook MJ. Multivariate correlates of adult blood pressures in nine North American populations: The Lipid Research Clinics Prevalence Study. Prev Med. 1982 Jul;11(4):391-402. doi: 10.1016/0091-7435(82)90043-3. No abstract available. PMID 7122431
- [Background] Sheffield LT, Haskell W, Heiss G, Kioschos M, Leon A, Roitman D, Schrott H: Safety of Exercise Testing Volunteer Subjects. The Lipid Research Clinics Prevalence Study Experience. J Cardiac Rehab 2(5):395-400, 1982
- [Background] Jacobs DR Jr, Barrett-Connor E. Retest reliability of plasma cholesterol and triglyceride. The Lipid Research Clinics Prevalence Study. Am J Epidemiol. 1982 Dec;116(6):878-85. doi: 10.1093/oxfordjournals.aje.a113490. PMID 7148814
- [Background] Rifkind BM, Heiss G, Tyroler HA, Williams OD: The Epidemiology of High Density Lipoproteins: The Lipid Research Clinics Program Prevalence Study. In: Proceedings of the Fourth International Meeting on Atherosclerosis - Atherosclerosis Clinical Evaluation and Therapy. Lenzi S, Descovich GC (Eds) Lancaster, England: MTP Press, Ltd., pp. 61-75, 1982
- [Background] Wahl PW, Walden CE, Knopp RH, Hoover JJ, Wallace RB, Rifkind BM: Effect of Estrogen/Progestin Potency on Lipid and Lipoprotein Cholesterol. The Lipid Research Clinics Program Prevalence Study. New Engl J Med 308:862-867, 1983
- [Background] Rifkind BM, Segal P. Lipid Research Clinics Program reference values for hyperlipidemia and hypolipidemia. JAMA. 1983 Oct 14;250(14):1869-72. PMID 6578354
- [Background] Criqui MH, Haskell WL, Heiss G, Tyroler HA, Green P, Rubenstein CJ. Predictors of systolic blood pressure response to treadmill exercise: the Lipid Research Clinics Program Prevalence Study. Circulation. 1983 Aug;68(2):225-33. doi: 10.1161/01.cir.68.2.225. PMID 6861301
- [Background] Greenberg RA, Green PP, Roggenkamp KJ, Barrett-Connor E, Tyroler HA, Heiss G. The constancy of parent-offspring similarity of total cholesterol throughout childhood and early adult life. The Lipid Research Clinics Program Prevalence Study. J Chronic Dis. 1984;37(11):833-8. doi: 10.1016/0021-9681(84)90016-x. PMID 6334097
- [Background] Green MS, Heiss G, Rifkind BM, Cooper GR, Williams OD, Tyroler HA. The ratio of plasma high-density lipoprotein cholesterol to total and low-density lipoprotein cholesterol: age-related changes and race and sex differences in selected North American populations. The Lipid Research Clinics Program Prevalence Study. Circulation. 1985 Jul;72(1):93-104. doi: 10.1161/01.cir.72.1.93. PMID 4006139
- [Background] Cowan LD, Wilcosky T, Criqui MH, Barrett-Connor E, Suchindran CM, Wallace R, Laskarzewski P, Walden C. Demographic, behavioral, biochemical, and dietary correlates of plasma triglycerides. Lipid Research Clinics Program Prevalence Study. Arteriosclerosis. 1985 Sep-Oct;5(5):466-80. doi: 10.1161/01.atv.5.5.466. PMID 4038160
- [Background] Barrett-Connor E, Wilcosky T, Wallace RB, Heiss G. Resting and exercise electrocardiographic abnormalities associated with sex hormone use in women. The Lipid Research Clinics Program Prevalence Study. Am J Epidemiol. 1986 Jan;123(1):81-8. doi: 10.1093/oxfordjournals.aje.a114226. PMID 3484419
- [Background] Knopp RH, Walden CE, Heiss G, Johnson JL, Wahl PW. Prevalence and clinical correlates of beta-migrating very-low-density lipoprotein. Lipid Research Clinics Program Prevalence Study. Am J Med. 1986 Sep;81(3):493-502. doi: 10.1016/0002-9343(86)90305-0. PMID 3463211
- [Background] Eisenberg S, Heiss G, Friedlander Y, Rifkind B, Segal P, Williams OD, Stein Y. Comparison of plasma lipids, lipoproteins and dyslipoproteinemia in Israel and the United States. The Lipid Research Clinics Program Prevalence Study. Atherosclerosis. 1986 Jan;59(1):63-74. doi: 10.1016/0021-9150(86)90034-1. PMID 3484958
- [Background] DeLong DM, DeLong ER, Wood PD, Lippel K, Rifkind BM. A comparison of methods for the estimation of plasma low- and very low-density lipoprotein cholesterol. The Lipid Research Clinics Prevalence Study. JAMA. 1986 Nov 7;256(17):2372-7. PMID 3464768
- [Background] Walden CE, Knopp RH, Johnson JL, Heiss G, Wahl PW, Hoover JJ. Effect of estrogen/progestin potency on clinical chemistry measures. The Lipid Research Clinics Program Prevalence Study. Am J Epidemiol. 1986 Mar;123(3):517-31. doi: 10.1093/oxfordjournals.aje.a114267. PMID 3946398
- [Background] Wilcosky T, Harris R, Weissfeld L. The prevalence and correlates of Rose Questionnaire angina among women and men in the Lipid Research Clinics Program Prevalence Study population. Am J Epidemiol. 1987 Mar;125(3):400-9. doi: 10.1093/oxfordjournals.aje.a114546. PMID 3812447
- [Background] Friedlander Y, Bucher KD, Namboodiri KK, Heiss G, Kark JD, Tyroler HA, Eisenberg S, Stein Y, Rifkind BM. Parent-offspring aggregation of plasma lipids in selected populations in North America and Israel. The Lipid Research Clinics Prevalence Study. Am J Epidemiol. 1987 Aug;126(2):268-79. doi: 10.1093/aje/126.2.268. PMID 3605055
- [Background] Wallace RB, Heiss G, Burrows B, Graves K. Contrasting diet and body mass among users and nonusers of oral contraceptives and exogenous estrogens: the Lipid Research Clinics Program Prevalence Study. Am J Epidemiol. 1987 May;125(5):854-9. doi: 10.1093/oxfordjournals.aje.a114601. PMID 3565359
- [Background] Kalsbeek WD, Kral KM, Wallace RB, Rifkind BM. Comparing mean levels of total cholesterol from visit 2 of the Lipid Research Clinics Prevalence Study with the second National Health and Nutrition Examination Survey. Am J Epidemiol. 1988 Nov;128(5):1038-53. doi: 10.1093/oxfordjournals.aje.a115048. PMID 3189280
- [Background] Ekelund LG, Suchindran CM, Karon JM, McMahon RP, Tyroler HA. Black-white differences in exercise blood pressure. The Lipid Research Clinics Program Prevalence Study. Circulation. 1990 May;81(5):1568-74. doi: 10.1161/01.cir.81.5.1568. PMID 2331768
- [Background] Tyroler HA. Epidemiology of plasma high-density lipoprotein cholesterol levels. The Lipid Research Clinics Program Prevalence Study. Introduction. Circulation. 1980 Nov;62(4 Pt 2):IV1-3. No abstract available. PMID 7418138
- [Background] Levy RI, Rifkind BM. The structure, function and metabolism of high-density lipoproteins: A status report. Circulation. 1980 Nov;62(4 Pt 2):IV4-8. PMID 6998596
- [Background] Albers JJ, Warnick GR, Johnson N, Bachorik PS, Muesing R, Lippel K, Williams OD. Quality control of plasma high-density lipoprotein cholesterol measurement methods. Circulation. 1980 Nov;62(4 Pt 2):IV9-18. No abstract available. PMID 7418148
- [Background] Williams OD, Mowery RL, Waldman GT. Common methods, different populations. The Lipid Research Clinics Program Prevalence Study. Circulation. 1980 Nov;62(4 Pt 2):IV18-23. PMID 7418141
- [Background] Davis CE, Gordon D, LaRosa J, Wood PD, Halperin M. Correlations of plasma high-density lipoprotein cholesterol levels with other plasma lipid and lipoprotein concentrations. Circulation. 1980 Nov;62(4 Pt 2):IV24-30. PMID 7188560
- [Background] Patten RL, Hewitt D, Waldman GT, Jones G, Little JA. Associations of plasma high-density lipoprotein cholesterol with clinical chemistry data. Circulation. 1980 Nov;62(4 Pt 2):IV31-41. PMID 7418142
- [Background] Ernst N, Fisher M, Smith W, Gordon T, Rifkind BM, Little JA, Mishkel MA, Williams OD. The association of plasma high-density lipoprotein cholesterol with dietary intake and alcohol consumption. The Lipid Research Clinics Prevalence Study. Circulation. 1980 Nov;62(4 Pt 2):IV41-52. PMID 7418143
- [Background] Haskell WL, Taylor HL, Wood PD, Schrott H, Heiss G. Strenuous physical activity, treadmill exercise test performance and plasma high-density lipoprotein cholesterol. The Lipid Research Clinics Program Prevalence Study. Circulation. 1980 Nov;62(4 Pt 2):IV53-61. PMID 7418144
- [Background] Glueck CJ, Taylor HL, Jacobs D, Morrison JA, Beaglehole R, Williams OD. Plasma high-density lipoprotein cholesterol: association with measurements of body mass. The Lipid Research Clinics Program Prevalence Study. Circulation. 1980 Nov;62(4 Pt 2):IV-62-9. PMID 7418145
- [Background] Criqui MH, Wallace RB, Heiss G, Mishkel M, Schonfeld G, Jones GT. Cigarette smoking and plasma high-density lipoprotein cholesterol. The Lipid Research Clinics Program Prevalence Study. Circulation. 1980 Nov;62(4 Pt 2):IV70-6. PMID 7418146
- [Background] Wallace RB, Hunninghake DB, Reiland S, Barrett-Connor E, Mackenthun A, Hoover J, Wahl P. Alterations of plasma high-density lipoprotein cholesterol levels associated with consumption of selected medications. The Lipid Research Clinics Program Prevalence Study. Circulation. 1980 Nov;62(4 Pt 2):IV77-82. PMID 6106533
- [Background] Beaglehole R, Trost DC, Tamir I, Kwiterovich P, Glueck CJ, Insull W, Christensen B. Plasma high-density lipoprotein cholesterol in children and young adults. The Lipid Research Clinics Program Prevalence Study. Circulation. 1980 Nov;62(4 Pt 2):IV83-92. PMID 7418147
- [Background] Halfon ST, Friedlander Y, Halperin G, Harlap S, Dennis BH, Moore MH, Mowery RL, Tyroler HA, Williams OD. Plasma high-density lipoprotein cholesterol, total cholesterol and triglyceride levels in 17-year-old Jewish residents of Jerusalem: a preliminary report. The Lipid Research Clinics Program Prevalence Study. Circulation. 1980 Nov;62(4 Pt 2):IV93-8. PMID 7418149
- [Background] Tyroler HA, Glueck CJ, Christensen B, Kwiterovich PO Jr. Plasma high-density lipoprotein cholesterol comparisons in black and white populations. The Lipid Research Clinics Program Prevalence Study. Circulation. 1980 Nov;62(4 Pt 2):IV99-107. PMID 7418150
- [Background] Heiss G, Haskell W, Mowery R, Criqui MH, Brockway M, Tyroler HA. Plasma high-density lipoprotein cholesterol and socioeconomic status. The Lipid Research Clinics Program Prevalence Study. Circulation. 1980 Nov;62(4 Pt 2):IV108-15. PMID 7418139
- [Background] Heiss G, Johnson NJ, Reiland S, Davis CE, Tyroler HA. The epidemiology of plasma high-density lipoprotein cholesterol levels. The Lipid Research Clinics Program Prevalence Study. Summary. Circulation. 1980 Nov;62(4 Pt 2):IV116-36. PMID 7418140
- [Background] Williams OD, Stinnett S, Chambless LE, Boyle KE, Bachorik PS, Albers JJ, Lippel K. Populations and methods for assessing dyslipoproteinemia and its correlates. The Lipid Research Clinics Program Prevalence Study. Circulation. 1986 Jan;73(1 Pt 2):I4-11. PMID 3940682
- [Background] LaRosa JC, Chambless LE, Criqui MH, Frantz ID, Glueck CJ, Heiss G, Morrison JA. Patterns of dyslipoproteinemia in selected North American populations. The Lipid Research Clinics Program Prevalence Study. Circulation. 1986 Jan;73(1 Pt 2):I12-29. PMID 3940679
- [Background] Kwiterovich PO Jr, Stewart P, Probstfield JL, Stinnett S, Chambless LE, Chase GA, Jacobs DR, Morrison JA. Detection of dyslipoproteinemia with the use of plasma total cholesterol and triglyceride as screening tests. The Lipid Research Clinics Program Prevalence Study. Circulation. 1986 Jan;73(1 Pt 2):I30-9. PMID 3940681
- [Background] Criqui MH, Cowan LD, Heiss G, Haskell WL, Laskarzewski PM, Chambless LE. Frequency and clustering of nonlipid coronary risk factors in dyslipoproteinemia. The Lipid Research Clinics Program Prevalence Study. Circulation. 1986 Jan;73(1 Pt 2):I40-50. PMID 3940683
- [Background] Glueck CJ, Laskarzewski PM, Suchindran CM, Chambless LE, Barrett-Connor E, Stewart P, Heiss G, Tyroler HA. Progeny's lipid and lipoprotein levels by parental mortality. The Lipid Research Clinics Program Prevalence Study. Circulation. 1986 Jan;73(1 Pt 2):I51-61. PMID 3940684
- [Background] Wallace RB, Pomrehn P, Heiss G, Chambless LE, Johnson N, Patten R, Lippel K, Rifkind BM. Alterations in clinical chemistry levels associated with the dyslipoproteinemias. The Lipid Research Clinics Program Prevalence Study. Circulation. 1986 Jan;73(1 Pt 2):I62-9. PMID 3940685
- [Background] Wallace RB, Hunninghake DB, Chambless LE, Heiss G, Wahl P, Barrett-Connor E. A screening survey of dyslipoproteinemias associated with prescription drug use. The Lipid Research Clinics Program Prevalence Study. Circulation. 1986 Jan;73(1 Pt 2):I70-9. PMID 2866852
- [Background] Little JA, Graves K, Suchindran CM, Milner J, McGuire V, Beaton G, Feather T, Mattson FH, Christiansen D, Williams OD. Customary diet, anthropometry, and dyslipoproteinemia in selected North American populations. The Lipid Research Clinics Program Prevalence Study. Circulation. 1986 Jan;73(1 Pt 2):I80-90. PMID 3940686
- [Background] Rubenstein C, Romhilt D, Segal P, Heiss G, Chambless LE, Boyle KE, Ekelund LG, Adolph R, Sheffield LT. Dyslipoproteinemias and manifestations of coronary heart disease. The Lipid Research Clinics Program Prevalence Study. Circulation. 1986 Jan;73(1 Pt 2):I91-9. PMID 3940687
- [Background] Pomrehn P, Duncan B, Weissfeld L, Wallace RB, Barnes R, Heiss G, Ekelund LG, Criqui MH, Johnson N, Chambless LE. The association of dyslipoproteinemia with symptoms and signs of peripheral arterial disease. The Lipid Research Clinics Program Prevalence Study. Circulation. 1986 Jan;73(1 Pt 2):I100-7. PMID 3940676
- [Background] Segal P, Insull W Jr, Chambless LE, Stinnett S, LaRosa JC, Weissfeld L, Halfon S, Kwiterovitch PO Jr, Little JA. The association of dyslipoproteinemia with corneal arcus and xanthelasma. The Lipid Research Clinics Program Prevalence Study. Circulation. 1986 Jan;73(1 Pt 2):I108-18. PMID 3940677
- [Background] Wilcosky TC, Kwiterovich PO Jr, Glueck CJ, Suchindran CM, Laskarzewski P, Christensen B, Tyroler HA. Dyslipoproteinemia in black participants. The Lipid Research Clinics Program Prevalence Study. Circulation. 1986 Jan;73(1 Pt 2):I119-25. PMID 3940678
- [Background] LaRosa JC, Levy RI, Hazzard WR. Some clinical implications of the results of the Lipid Research Clinics Program Prevalence Study. Circulation. 1986 Jan;73(1 Pt 2):I126-33. No abstract available. PMID 3940680
- [Background] US-USSR Steering Committee for Problem Area 1: A Comparison of High Blood Pressure Prevalence and Treatment Status in Selected US and USSR Populations. The Pathogenesis of Atherosclerosis. In: First Joint US-USSR Symposium on Hypertension, Sochi, USSR, U.S. Department of Health, Education, and Welfare, NIH Publication No. 79-1272, 432-433, August, 1979
- [Background] Lipid Research Clinics Program: Protocol of the Lipid Research Clinics Program Prevalence Study. Central Patient Registry and Coordinating Center, Department of Biostatistics, University of North Carolina at Chapel Hill, 1974
- [Background] Central Patient Registry and Coordinating Center for the Lipid Research Clinics: Reference Manual for the Lipid Research Clinics Prevalence Study, vols. 1 and 2. Chapel Hill, Department of Biostatistics, University of North Carolina, February 1974
- [Background] Lipid Research Clinics Program: Manual of Laboratory Operations, vol. 1. Lipid and Lipoprotein Analysis. Washington, DC., U.S. Government Printing Office, DHEW Publication No. (NIH) 75-628, May 1974
- [Background] Wallace RB, Hoover J, Sandler D, Rifking BM, Tyroler HA. Altered plasma-lipids associated with oral contraceptive or oestrogen consumption. The Lipid Research Clinic Program. Lancet. 1977 Jul 2;2(8027):11-4. doi: 10.1016/s0140-6736(77)90005-8. PMID 69101
- [Background] Rifkind BM, Tamir I, Heiss G.: Preliminary High-Density Lipoprotein Findings: The Lipid Research Clinics Program. In: Gotto AM, Jr. Miller NE, Oliver MF, (Eds), High Density Lipoproteins and Atherosclerosis. Amsterdam: Elsevier/North Holland Biomedical press, pp. 109-119, 1978
- [Background] Rifkind BM, Tamir I, Heiss G, Wallace RB, Tyroler HA. Distribution of high density and other lipoproteins in selected LRC prevalence study populations: a brief survey. Lipids. 1979 Jan;14(1):105-12. doi: 10.1007/BF02533578. PMID 218067
- [Background] Beaglehole R, LaRosa JC, Heiss G, Davis CE, Williams OD, Tyroler HA, Rifkind BM. Serum cholesterol, diet, and the decline in coronary heart disease mortality. Prev Med. 1979 Sep;8(5):538-47. doi: 10.1016/0091-7435(79)90329-3. No abstract available. PMID 504077
- [Background] Wallace RB, Tamir I, Heiss G, Rifkind BM, Christensen B, Glueck CJ. Plasma lipids, lipoproteins, and blood pressure in female adolescents using oral contraceptives. J Pediatr. 1979 Dec;95(6):1055-9. doi: 10.1016/s0022-3476(79)80311-x. PMID 501486
- [Background] Wallace RB, Hoover J, Barrett-Connor E, Rifkind BM, Hunninghake DB, Mackenthun A, Heiss G. Altered plasma lipid and lipoprotein levels associated with oral contraceptive and oestrogen use. Report from the Medications Working Group of the Lipid Research Clinics Program. Lancet. 1979 Jul 21;2(8134):112-5. PMID 88553
- [Background] Plasma lipid distributions in selected North American populations: the Lipid Research Clinics Program Prevalence Study. The Lipid Research Clinics Program Epidemiology Committee. Circulation. 1979 Aug;60(2):427-39. doi: 10.1161/01.cir.60.2.427. PMID 312704
- [Background] Heiss G, Tamir I, Davis CE, Tyroler HA, Rifkand BM, Schonfeld G, Jacobs D, Frantz ID Jr. Lipoprotein-cholesterol distributions in selected North American populations: the lipid research clinics program prevalence study. Circulation. 1980 Feb;61(2):302-15. doi: 10.1161/01.cir.61.2.302. No abstract available. PMID 7351055
- [Background] The Lipid Research Clinics Population Studies Data Book. Volume I. The Prevalence Study. U.S. Department of Health and Human Services. NIH Publication No. 80-1527, July 1980
- [Background] Rifkind BM, LaRosa J. Heiss G: The Prevalence of Hyperlipidemia in Selected North American Populations. In: Atherosclerosis V. Proceedings of the Fifth International Symposium on Atherosclerosis (Gotto AM, Ed) New York:Springer-Verlag, pp. 264-267; 829-830, 1980
- [Background] US-USSR Steering Committee for Problem Area 1: US-USSR First Lipoprotein Symposium. Laboratory Research Joint Population Studies, Leningrad, USSR. The Pathogenesis of Atherosclerosis. U.S. Department of Health and Human Services. NIH Publication No. 83-1966, November 1982
- [Background] Williams OD, Rywik SL, Tyroler HA, Sznajd J, McClish DK, Ingram D, Maciolowski M: The U.S. - Polish Pilot Study. In: USA-Poland Symposium, Ischemic Heart Disease. U.S. Department of Health and Human Services. NIH Publication No. 82-1273, pp. 1-8 March 1982
- [Background] Nutrient intake and its association with high-density lipoprotein and low-density lipoprotein cholesterol in selected US and USSR subpopulations. The US-USSR Steering Committee for Problem Area I: The pathogenesis of atherosclerosis. Am J Clin Nutr. 1984 Jun;39(6):942-52. doi: 10.1093/ajcn/39.6.942. PMID 6609630
- [Background] Ingram DD, Thorn MD, Stinnett SS, Deev AD. U.S.S.R. and U.S. nutrient intake, plasma lipids, and lipoproteins in men ages 40-59 sampled from Lipid Research Clinics populations. Prev Med. 1985 May;14(3):264-71. doi: 10.1016/0091-7435(85)90055-6. PMID 4059187
- [Background] The Lipid Research Clinics Population Studies Data Book. Volume III. The USSR First Prevalence Study. US Department of Health and Human Services. NIH Publication No.87-2727, November 1986
- [Background] Abernathy JR, Thorn MD, Trobaugh GB, Ekelund LG, Maciolowski M, Lupovetsky B, Shelnova S, Zhukovsky G, Shestov D, Deev A. Prevalence of ischemic resting and stress electrocardiographic abnormalities and angina among 40- to 59-year-old men in selected U.S. and U.S.S.R. populations. Circulation. 1988 Feb;77(2):270-8. doi: 10.1161/01.cir.77.2.270. PMID 3338123
- [Background] Abernathy JR, Thorn MD, Ekelund LG, Holme I, Stinnett SS, Shestov DB, Deev AD. Correlates of systolic and diastolic blood pressure in men 40 to 59 years of age sampled from United States of America and Union of Soviet Socialist Republics Lipid Research Clinics populations. Am J Cardiol. 1988 May 1;61(13):1071-5. doi: 10.1016/0002-9149(88)90128-2. PMID 3259070
- [Background] The Lipid Research Clinics Population Studies Data Book. Volume IV. The USSR Second Prevalence Study. US Department of Health and Human Services. NIH Publication No.90-2995, June 1990
- [Background] Tyroler HA. The lipid research clinics population-based family study. Prog Clin Biol Res. 1979;32:647-52. No abstract available. PMID 523489
- [Background] Segal P, Rifkind BM, Schull WJ. Genetic factors in lipoprotein variation. Epidemiol Rev. 1982;4:137-60. doi: 10.1093/oxfordjournals.epirev.a036244. No abstract available. PMID 6754405
- [Background] Karlin S, Williams PT, Farquhar JW, Barrett-Connor E, Hoover J, Wahl PW, Haskell WL, Bergelin RO, Suarez L. Association arrays for the study of familial height, weight, lipid, and lipoprotein similarity in three West Coast populations. Am J Epidemiol. 1982 Dec;116(6):1001-21. doi: 10.1093/oxfordjournals.aje.a113485. PMID 7148811
- [Background] Morrison JA, Namboodiri K, Green P, Martin J, Glueck CJ. Familial aggregation of lipids and lipoproteins and early identification of dyslipoproteinemia. The Collaborative Lipid Research Clinics Family Study. JAMA. 1983 Oct 14;250(14):1860-8. PMID 6620483
- [Background] Namboodiri KK, Green PP, Kaplan EB, Tyroler HA, Morrison JA, Chase GA, Elston RC, Rifkind BM, Glueck CJ. Family aggregation of high density lipoprotein cholesterol. Collaborative lipid research clinics program family study. Arteriosclerosis. 1983 Nov-Dec;3(6):616-26. doi: 10.1161/01.atv.3.6.616. PMID 6651617
- [Background] The Collaborative Lipid Research Clinics Program Family Study. I. Study design and description of data. Am J Epidemiol. 1984 Jun;119(6):931-43. PMID 6731432
- [Background] Namboodiri KK, Green PP, Walden C, Kaplan EB, Dawson D, Kelly K, Maciolowski M, Morrison JA, Elston RC, Austin M, et al. The Collaborative Lipid Research Clinics Program Family Study. II. Response rates, representativeness of the sample, and stability of lipid and lipoprotein levels. Am J Epidemiol. 1984 Jun;119(6):944-58. doi: 10.1093/oxfordjournals.aje.a113816. PMID 6731433
- [Background] Green PP, Namboodiri KK, Hannan P, Martin J, Owen AR, Chase GA, Kaplan EB, Williams L, Elston RC. The Collaborative Lipid Research Clinics Program Family Study. III. Transformations and covariate adjustments of lipid and lipoprotein levels. Am J Epidemiol. 1984 Jun;119(6):959-74. doi: 10.1093/oxfordjournals.aje.a113817. PMID 6731434
- [Background] Namboodiri KK, Green PP, Kaplan EB, Morrison JA, Chase GA, Elston RC, Owen AR, Rifkind BM, Glueck CJ, Tyroler HA. The Collaborative Lipid Research Clinics Program Family Study. IV. Familial associations of plasma lipids and lipoproteins. Am J Epidemiol. 1984 Jun;119(6):975-96. doi: 10.1093/oxfordjournals.aje.a113818. PMID 6731435
- [Background] Green P, Owen AR, Namboodiri K, Hewitt D, Williams LR, Elston RC. The Collaborative Lipid Research Clinics Program Family Study: detection of major genes influencing lipid levels by examination of heterogeneity of familial variances. Genet Epidemiol. 1984;1(2):123-41. doi: 10.1002/gepi.1370010204. PMID 6544235
- [Background] Namboodiri KK, Kaplan EB, Heuch I, Elston RC, Green PP, Rao DC, Laskarzewski P, Glueck CJ, Rifkind BM. The Collaborative Lipid Research Clinics Family Study: biological and cultural determinants of familial resemblance for plasma lipids and lipoproteins. Genet Epidemiol. 1985;2(3):227-54. doi: 10.1002/gepi.1370020302. PMID 4054601
- [Background] Heuch I, Namboodiri KK, Green PP, Kaplan EB, Laskarzewski P, Glueck CJ, Elston RC. A multivariate analysis of familial associations of lipoprotein levels in the Lipid Research Clinics Collaborative Family Study: I. Familial correlation and regression analyses. Genet Epidemiol. 1985;2(3):283-300. doi: 10.1002/gepi.1370020306. PMID 3863779
- [Background] Bucher KD, Kaplan EB, Namboodiri KK, Glueck CJ, Laskarzewski P, Rifkind BM. Segregation analysis of low levels of high-density lipoprotein cholesterol in the collaborative Lipid Research Clinics Program Family Study. Am J Hum Genet. 1987 Jun;40(6):489-502. PMID 3591798
- [Background] Bucher KD, Friedlander Y, Kaplan EB, Namboodiri KK, Kark JD, Eisenberg S, Stein Y, Rifkind BM. Biological and cultural sources of familial resemblance in plasma lipids: a comparison between North America and Israel--the Lipid Research Clinics Program. Genet Epidemiol. 1988;5(1):17-33. doi: 10.1002/gepi.1370050103. PMID 3360301
- [Background] Bush TL, Cowan LD, Barrett-Connor E, Criqui MH, Karon JM, Wallace RB, Tyroler HA, Rifkind BM. Estrogen use and all-cause mortality. Preliminary results from the Lipid Research Clinics Program Follow-Up Study. JAMA. 1983 Feb 18;249(7):903-6. doi: 10.1001/jama.249.7.903. PMID 6823043
- [Background] Gordon DJ, Ekelund LG, Karon JM, Probstfield JL, Rubenstein C, Sheffield LT, Weissfeld L. Predictive value of the exercise tolerance test for mortality in North American men: the Lipid Research Clinics Mortality Follow-up Study. Circulation. 1986 Aug;74(2):252-61. doi: 10.1161/01.cir.74.2.252. PMID 3731417
- [Background] Criqui MH, Cowan LD, Tyroler HA, Bangdiwala S, Heiss G, Wallace RB, Cohn R. Lipoproteins as mediators for the effects of alcohol consumption and cigarette smoking on cardiovascular mortality: results form the Lipid Research Clinics Follow-up Study. Am J Epidemiol. 1987 Oct;126(4):629-37. doi: 10.1093/oxfordjournals.aje.a114702. PMID 3631053
- [Background] Bush TL, Barrett-Connor E, Cowan LD, Criqui MH, Wallace RB, Suchindran CM, Tyroler HA, Rifkind BM. Cardiovascular mortality and noncontraceptive use of estrogen in women: results from the Lipid Research Clinics Program Follow-up Study. Circulation. 1987 Jun;75(6):1102-9. doi: 10.1161/01.cir.75.6.1102. PMID 3568321
- [Background] Ekelund LG, Haskell WL, Johnson JL, Whaley FS, Criqui MH, Sheps DS. Physical fitness as a predictor of cardiovascular mortality in asymptomatic North American men. The Lipid Research Clinics Mortality Follow-up Study. N Engl J Med. 1988 Nov 24;319(21):1379-84. doi: 10.1056/NEJM198811243192104. PMID 3185648
- [Background] Gordon DJ, Probstfield JL, Garrison RJ, Neaton JD, Castelli WP, Knoke JD, Jacobs DR Jr, Bangdiwala S, Tyroler HA. High-density lipoprotein cholesterol and cardiovascular disease. Four prospective American studies. Circulation. 1989 Jan;79(1):8-15. doi: 10.1161/01.cir.79.1.8. PMID 2642759
- [Background] Bangdiwala SI, Cohn R, Hazard C, Davis CE, Prineas RJ. Comparisons of cause of death verification methods and costs in the lipid research clinics program mortality follow-up study. Control Clin Trials. 1989 Jun;10(2):167-87. doi: 10.1016/0197-2456(89)90029-9. PMID 2666025
- [Background] Wilcosky T, Hyde J, Anderson JJ, Bangdiwala S, Duncan B. Obesity and mortality in the Lipid Research Clinics Program Follow-up Study. J Clin Epidemiol. 1990;43(8):743-52. doi: 10.1016/0895-4356(90)90232-e. PMID 2384763
- [Background] Jacobs DR Jr, Mebane IL, Bangdiwala SI, Criqui MH, Tyroler HA. High density lipoprotein cholesterol as a predictor of cardiovascular disease mortality in men and women: the follow-up study of the Lipid Research Clinics Prevalence Study. Am J Epidemiol. 1990 Jan;131(1):32-47. doi: 10.1093/oxfordjournals.aje.a115483. PMID 2293751
- [Background] Cowan LD, O'Connell DL, Criqui MH, Barrett-Connor E, Bush TL, Wallace RB. Cancer mortality and lipid and lipoprotein levels. Lipid Research Clinics Program Mortality Follow-up Study. Am J Epidemiol. 1990 Mar;131(3):468-82. doi: 10.1093/oxfordjournals.aje.a115521. PMID 2301356
- [Background] Pekkanen J, Linn S, Heiss G, Suchindran CM, Leon A, Rifkind BM, Tyroler HA. Ten-year mortality from cardiovascular disease in relation to cholesterol level among men with and without preexisting cardiovascular disease. N Engl J Med. 1990 Jun 14;322(24):1700-7. doi: 10.1056/NEJM199006143222403. PMID 2342536
- [Background] Williams OD, Heiss G, Beaglehole R, Dennis B, Bazzarre T, Tyroler HA: Hyperlipidemia and Nutrition: Data Base and Trends. Atherosclerosis Reviews 7:145-156, 1980
- [Background] Dennis B, Ernst N, Hjortland M, Tillotson J, Grambsch V. The NHLBI nutrition data system. J Am Diet Assoc. 1980 Dec;77(6):641-7. PMID 6893713
- [Background] Beaton GH, Milner J, Corey P, McGuire V, Cousins M, Stewart E, de Ramos M, Hewitt D, Grambsch PV, Kassim N, Little JA. Sources of variance in 24-hour dietary recall data: implications for nutrition study design and interpretation. Am J Clin Nutr. 1979 Dec;32(12):2546-59. doi: 10.1093/ajcn/32.12.2546. No abstract available. PMID 506977
- [Background] Report of the Evaluation Panels for the NHLBI Dietary Data Collection System. (Unpublished report, available in limited quantities from the Lipid Metabolism Branch, NHLBI), 0000
- [Background] Gordon T, Fisher M, Rifkind BM. Some difficulties inherent in the interpretation of dietary data from free-living populations. Am J Clin Nutr. 1984 Jan;39(1):152-6. doi: 10.1093/ajcn/39.1.152. PMID 6606975
- [Background] Brewer ER, Kassim N, Cronin FJ, Dennis BH, Kuczmarski RJ, Haynes S, Graves K. Food group system of analysis with special attention to type and amount of fat--methodology. J Am Diet Assoc. 1987 May;87(5):584-92. PMID 3571775
- [Background] Rifkind BM. Nutrient--high-density lipoprotein relationships: an overview. Prog Biochem Pharmacol. 1983;19:89-109. No abstract available. PMID 6338526
- [Background] Salz KM, Tamir I, Ernst N, Kwiterovich P, Glueck C, Christensen B, Larsen R, Pirhonen D, Prewitt TE, Scott LW. Selected nutrient intakes of free-living white children ages 6-19 years. The Lipid Research Clinics Program Prevalence Study. Pediatr Res. 1983 Feb;17(2):124-30. doi: 10.1203/00006450-198302000-00009. PMID 6828330
- [Background] Glueck CJ, Waldman G, McClish DK, Morrison JA, Khoury P, Larsen R, Salz K, Rifkind BM, Mattson FH. Relationships of nutrient intake to lipids and lipoproteins in 1234 white children. The Lipid Research Clinics Prevalence Study. Arteriosclerosis. 1982 Nov-Dec;2(6):523-36. doi: 10.1161/01.atv.2.6.523. PMID 7181737
- [Background] Gordon T, Fisher M, Ernst N, Rifkind BM. Relation of diet to LDL cholesterol, VLDL cholesterol, and plasma total cholesterol and triglycerides in white adults. The Lipid Research Clinics Prevalence Study. Arteriosclerosis. 1982 Nov-Dec;2(6):502-12. doi: 10.1161/01.atv.2.6.502. PMID 6983876
- [Background] Gordon DJ, Salz KM, Roggenkamp KJ, Franklin FA Jr. Dietary determinants of plasma cholesterol change in the recruitment phase of the Lipid Research Clinics Coronary Primary Prevention Trial. Arteriosclerosis. 1982 Nov-Dec;2(6):537-48. doi: 10.1161/01.atv.2.6.537. PMID 7181738
- [Background] Schwarz W, Trost DC, Reiland SL, Rifkind BM, Heiss G. Correlates of low density lipoprotein cholesterol: associations with physical, chemical, dietary, and behavioral characteristics. Arteriosclerosis. 1982 Nov-Dec;2(6):513-22. doi: 10.1161/01.atv.2.6.513. PMID 6983877
- [Background] The Lipid Research Clinics Population Studies Data Book. Volume II. The Prevalence Study - Nutrient Intake. U.S. Department of Health and Human Services. NIH Publication No. 82-2014, September 1982
- [Background] Goor R, Hosking JD, Dennis BH, Graves KL, Waldman GT, Haynes SG. Nutrient intakes among selected North American populations in the Lipid Research Clinics Prevalence Study: composition of fat intake. Am J Clin Nutr. 1985 Feb;41(2):299-311. doi: 10.1093/ajcn/41.2.299. PMID 3969938
- [Background] Dennis BH, Haynes SG, Anderson JJ, Liu-Chi SB, Hosking JD, Rifkind BM. Nutrient intakes among selected North American populations in the Lipid Research Clinics Prevalence Study: composition of energy intake. Am J Clin Nutr. 1985 Feb;41(2):312-29. doi: 10.1093/ajcn/41.2.312. PMID 3969939
- [Background] Fisher M, Gordon T. The relation of drinking and smoking habits to diet: the Lipid Research Clinics Prevalence Study. Am J Clin Nutr. 1985 Mar;41(3):623-30. doi: 10.1093/ajcn/41.3.623. PMID 3976562
- [Background] Kaufmann NA, Dennis BH, Heiss G, Friedlander Y, Kark JD, Stein Y. Comparison of nutrient intakes of selected populations in the United States and Israel: the Lipid Research Clinics prevalence study. Am J Clin Nutr. 1986 Apr;43(4):604-20. doi: 10.1093/ajcn/43.4.604. PMID 3962910
- [Background] Kuczmarski RJ, Brewer ER, Cronin FJ, Dennis B, Graves K, Haynes S. Food choices among white adolescents: the Lipid Research Clinics Prevalence Study. Pediatr Res. 1986 Apr;20(4):309-15. doi: 10.1203/00006450-198604000-00006. PMID 3703620
- [Background] Prewitt TE, Haynes SG, Graves K, Haines PS, Tyroler HA. Nutrient intake, lipids, and lipoprotein cholesterols in black and white children: the Lipid Research Clinics Prevalence Study. Prev Med. 1988 May;17(3):247-62. doi: 10.1016/0091-7435(88)90001-1. PMID 3405982
- [Background] Manual of Laboratory Operations: LRC Program, Vol. 1: Lipid and Lipoprotein Analysis. DHEW Publication No. (NIH) 75-628. May 1974. Revised version issued October, 1982
- [Background] Bachorik PS, Wood PD, Albers JJ, Steiner P, Dempsey M, Kuba K, Warnick R, Karlsson L. Plasma high-density lipoprotein cholesterol concentrations determined after removal of other lipoproteins by heparin/manganese precipitation or by ultracentrifugation. Clin Chem. 1976 Nov;22(11):1828-34. PMID 184986
- [Background] Cholesterol and triglyceride concentrations in serum/plasma pairs. Clin Chem. 1977 Jan;23(1):60-3. PMID 832373
- [Background] Lippel K, Ahmed S, Albers JJ, Bachorik P, Cooper G, Helms R, Williams J. Analytical performance and comparability of the determination of cholesterol by 12 Lipid-Research Clinics. Clin Chem. 1977 Sep;23(9):1744-52. PMID 890919
- [Background] Ahmed S, Lippel K, Bachorik P, Albers J, Williams J, Cooper G. Analytical performance and comparability of the determination of triglycerides by 12 Lipid Research Clinic laboratories. Clin Chem. 1978 Feb;24(2):330-8. PMID 627065
- [Background] Bachorik PS, Cooper G, Lippel K, and Ahmed S: Standardization of Cholesterol and Triglyceride Measurements by 12 Lipid Research Clinics. In Protides of the Biological Fluids (Proceedings of the 25th Colloquium), H. Peeters, (Ed). New York: Pergamon Press, pp. 307-314, 1978
- [Background] Albers JJ, Warnick GR, Wiebe D, King P, Steiner P, Smith L, Breckenridge C, Chow A, Kuba K, Weidman S, Arnett H, Wood P, Shlagenhaft A. Multi-laboratory comparison of three heparin-Mn2+ precipitation procedures for estimating cholesterol in high-density lipoprotein. Clin Chem. 1978 Jun;24(6):853-6. PMID 207461
- [Background] Lippel K, Ahmed S, Albers JJ, Bachorik P, Muesing R, Winn C. External quality-control survey of cholesterol analyses performed by 12 lipid research clinics. Clin Chem. 1978 Sep;24(9):1477-84. PMID 688605
- [Background] Shalnova S, Shestov DB, Ekelund LG, Abernathy JR, Plavinskaya S, Thomas RP, Williams DH, Deev A, Davis CE. Blood pressure and heart rate response during exercise in men and women in the USA and Russia lipid research clinics prevalence study. Atherosclerosis. 1996 Apr 26;122(1):47-57. doi: 10.1016/0021-9150(95)05746-3. PMID 8724111
- [Background] Collaborative US-USSR study on the prevalence of dyslipoproteinemias and ischemic heart disease in American and Soviet populations. Prepared by the US-USSR Steering Committee for Problem Area 1: the pathogenesis of atherosclerosis. Am J Cardiol. 1977 Aug;40(2):260-8. doi: 10.1016/0002-9149(77)90017-0. PMID 195454
- [Background] Esrey KL, Joseph L, Grover SA. Relationship between dietary intake and coronary heart disease mortality: lipid research clinics prevalence follow-up study. J Clin Epidemiol. 1996 Feb;49(2):211-6. doi: 10.1016/0895-4356(95)00066-6. PMID 8606322
- [Background] Mora S, Redberg RF, Cui Y, Whiteman MK, Flaws JA, Sharrett AR, Blumenthal RS. Ability of exercise testing to predict cardiovascular and all-cause death in asymptomatic women: a 20-year follow-up of the lipid research clinics prevalence study. JAMA. 2003 Sep 24;290(12):1600-7. doi: 10.1001/jama.290.12.1600. PMID 14506119
- Available data/document: Individual Participant Data Set: LRC-PS — http://biolincc.nhlbi.nih.gov/studies/lrcps/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/lrcps/